



# **CLINICAL PERFORMANCE STUDY PLAN**

## EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test

### AnteoTech LTD.

Document reference number: Version 3.0

Date: 19-Sep-2022

Template CA-06.17.02-A 



AnteoTech LTD.
EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test
Clinical Performance Study
CPSP Ver 3.0, 19Sep2022

#### **CONTACT INFORMATION**

#### SPONSOR AND LEGAL MANUFACTURER

AnteoTech Ltd Unit 4, 26 Brandl Street Brisbane Technology Park Eight Mile Plains QLD 4113 Australia

#### **AUTHORIZED REPRESENTATIVE IN EU:**

MT Promedt Consulting GmbH Altenhofstrasse 80 66386 St. Ingbert Germany

CRO:
AKRN Scientific Consulting

INVESTIGATIONAL SITE (S):




#### **CLINICAL PERFORMANCE STUDY PLAN (CPSP) SUMMARY**

| Version Number | 3.0 |
|---|---|
| Date | 19-Sep-2022 |
| Sponsor | AnteoTech Ltd Unit 4, 26 Brandl Street Brisbane Technology Park Eight Mile Plains QLD 4113 Australia EU authorized representative: MT Promedt Consulting GmbH Altenhofstrasse 80 66386 St. Ingbert Germany |
| Clinical Performance<br>Study Name | EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test Clinical Performance Study |
| Clinical Performance<br>Study Code | |
| Objectives | To determine the diagnostic accuracy in terms of specificity and sensitivity of the EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test in the diagnosis of SARS-CoV-2 in specimens prospectively collected by healthcare professionals from subjects suspected of COVID-19 disease or with unknown COVID-19 status. |
| Device Under<br>Investigation | EuGeni SARS-CoV-2 Ag RDT assay and EuGeni Reader |
| Number of Required<br>Specimens | A minimum estimated of 1850 prospective specimens divided as follows: Nasopharyngeal specimen collection: 300 positive specimens from symptomatic subjects 120 negative specimens from hospitalized patients 505 negative specimens from subjects with respiratory symptoms Combined nasal mid-turbinate and throat specimen collection: 300 positive specimens from symptomatic subjects 120 negative specimens from hospitalized patients 505 negative specimens from subjects with respiratory symptoms |
| Planned Number of<br>Sites | Up to 10 sites in Europe |
| Study Design | This is a non-interventional, two-arm, prospective, non-randomized, open-label and multi-center Clinical Performance Study |




| · | Ť. |
|---|---|
| | To assess the EuGeni SARS-CoV-2 Ag RDT diagnostic accuracy in terms of sensitivity and specificity measured as the following: |
| Primary Endpoints | <ul> <li>The diagnostic sensitivity will be assessed as the ability to identify the presence of a target marker associated with SARS-CoV-2, of nasopharyngeal specimens and combined nasal mid-turbinate and throat specimens, respectively, compared with gold-standard SARS-CoV-2 RT-PCR.</li> <li>The diagnostic specificity will be assessed as the ability to recognise the absence of a target marker associated with SARS CoV-2, of nasopharyngeal specimens and combined nasal mid-turbinate and throat specimens, respectively, compared with gold-standard SARS-</li> </ul> |
| | CoV-2 RT-PCR. |
| Secondary Endpoint | To compare the specificity and sensitivity rates of EuGeni SARS-CoV-2 Ag RDT between the two specimen collection methods. |
| | <ol> <li>Specimens from subjects over 12 years old agreeing to participate in the<br/>study and with a legal representative able to provide informed consent,<br/>OR;</li> </ol> |
| Inclusion Criteria | <ol><li>Specimens from subjects over 18 years old able to provide informed<br/>consent.</li></ol> |
| | <ol> <li>Specimens collected with nasopharyngeal swabs, OR;</li> <li>Combined nasal mid-turbinate and throat specimen collection.</li> </ol> |
| | <ol> <li>Specimens and testing methods that are not deemed to be in line with<br/>gold-standard RT-PCR standards.</li> </ol> |
| | <ol><li>Specimens stored for over 2 hours at 2-8 °C temperature between<br/>collection and testing with EuGeni SARS-CoV-2 Ag RDT</li></ol> |
| Exclusion Criteria | <ol><li>Specimens stored for over 5 days at -20°C between collection and<br/>testing with RT-PCR.</li></ol> |
| | <ol> <li>Specimens stored for over 24h at 4°C between collection and testing<br/>with RT-PCR.</li> </ol> |
| | <ol><li>Contamination and/or deterioration of the specimen which, in the opinion<br/>of the investigator, may affect its handling and/or analysis.</li></ol> |
| | <ol><li>The subject is deemed unsuitable to participate in the study by the<br/>investigator.</li></ol> |
| Coordinating<br>Investigator | |
| Electronic Data<br>Capture (EDC) | |
| Data Management & Biostatistics | |
| Contract Research<br>Organization (CRO) | AKRN Scientific Consulting S.L. (Madrid, Spain) |
| Expected Duration of the Study | |




AnteoTech LTD. EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test Clinical Performance Study CPSP Ver 3.0, 19Sep2022

| <u> </u> |
|----------|

Investigational Site Name





| ) |
|---|
| 8 |






| <br> |
|-----------------|
| <br><del></del> |




AnteoTech LTD.
EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test
Clinical Performance Study
CPSP Ver 3.0, 19Sep2022

#### **COMPLIANCE STATEMENT:**

This clinical performance study will be conducted in accordance with this Clinical Performance Study Plan, the Declaration of Helsinki, law 14/2007 of 3 July 2007 on Biomedical Research, applicable Good Clinical Practices, ISO 20916:2019 standards and regulations: EU 2017/746 of the European Parliament and of the Council of 5 April 2017 on in vitro diagnostic medical devices (IVDR), repealing Directive 98/79/EC and Commission Decision 2010/227/EU, EU General Data Protection Regulation and WHO International health regulations.

The most stringent requirements, guidelines or regulations must always be followed. The conduct of the clinical performance study will be approved by the appropriate Institutional Review Board (IRB)/Ethics Committee (EC) of the respective investigational site and by the applicable regulatory authorities.

#### CONFIDENTIALITY STATEMENT

This document is confidential and is to be distributed for review only to investigators, potential investigators, consultants, study staff, and applicable independent Ethics Committees or Competent Authorities. The contents of this document shall not be disclosed to others without written authorization from the Sponsor unless it is necessary to obtain informed consent from potential study participants.

Template CA-06.17.02-A 



#### **TABLE OF CONTENTS**

| 1. | INTRODUCTION | 12 |
|---|---|---|
| 1.1 | BACKGROUND AND RATIONALE | 12 |
| 2. | IN-VITRO DIAGNOSTIC MEDICAL DEVICE OVERVIEW | 13 |
| 2.1 | IVD MEDICAL DEVICE UNDER INVESTIGATION | 13 |
| 2.2 | INTENDED PURPOSE | 13 |
| 2.3 | INTENDED USER | 14 |
| 2.4 | MECHANISM OF ACTION OF THE DEVICE UNDER INVESTIGATION | 14 |
| 2.5 | DEVICE HANDLING | 14 |
| 3. | CLINICAL PERFORMANCE STUDY OVERVIEW | 15 |
| 3.1 | CLINICAL PERFORMANCE STUDY OBJECTIVE | 15 |
| 4. | CLINICAL PERFORMANCE STUDY DESIGN AND PROCEDURES | 16 |
| 4.1 | CLINICAL PERFORMANCE STUDY DESIGN | 16 |
| 4.2 | CLINICAL PERFORMANCE STUDY PROCEDURES | 16 |
| | 4.2.1 Informed Consent and Specimen collection | |
| | 4.2.2.1 Specimen handling and storage | |
| 4.3 | MEASURES TAKEN TO AVOID AND MINIMIZE BIAS | |
| 4.3<br>5. | MEASURES TAKEN TO AVOID AND MINIMIZE BIAS ENDPOINTS | |
| | | 19 |
| 5. | ENDPOINTS | 19<br>19 |
| 5.<br>5.1 | PRIMARY ENDPOINTS | 19<br>19<br>19 |
| 5.<br>5.1<br>5.2 | PRIMARY ENDPOINTS | 19<br>19<br>19<br>20 |
| 5.<br>5.1<br>5.2<br>6. | PRIMARY ENDPOINTS | 19<br>19<br>19<br>20<br>20 |
| 5.<br>5.1<br>5.2<br>6. | ENDPOINTS PRIMARY ENDPOINTS SECONDARY ENDPOINT SELECTION OF SPECIMENS SPECIMENS AND SUBJECTS PROVIDING SPECIMENS 6.1.1 Subject Screening 6.1.2 Informed Consent | 19<br>19<br>19<br>20<br>20<br>20 |
| 5.<br>5.1<br>5.2<br>6.<br>6.1 | ENDPOINTS PRIMARY ENDPOINTS SECONDARY ENDPOINT SELECTION OF SPECIMENS SPECIMENS AND SUBJECTS PROVIDING SPECIMENS 6.1.1 Subject Screening 6.1.2 Informed Consent 6.1.2.1 Special Circumstances for Informed Consent | 19<br>19<br>19<br>20<br>20<br>20<br>20<br>21 |
| 5.<br>5.1<br>5.2<br>6.<br>6.1 | ENDPOINTS PRIMARY ENDPOINTS SECONDARY ENDPOINT SELECTION OF SPECIMENS SPECIMENS AND SUBJECTS PROVIDING SPECIMENS 6.1.1 Subject Screening 6.1.2 Informed Consent 6.1.2.1 Special Circumstances for Informed Consent ELIGIBILITY CRITERIA | 19<br>19<br>20<br>20<br>20<br>21<br>21 |
| 5.<br>5.1<br>5.2<br>6.<br>6.1 | ENDPOINTS PRIMARY ENDPOINTS SECONDARY ENDPOINT SELECTION OF SPECIMENS SPECIMENS AND SUBJECTS PROVIDING SPECIMENS 6.1.1 Subject Screening 6.1.2 Informed Consent 6.1.2.1 Special Circumstances for Informed Consent | 19<br>19<br>20<br>20<br>20<br>21<br>21<br>21 |
| 5.<br>5.1<br>5.2<br>6.<br>6.1 | ENDPOINTS PRIMARY ENDPOINTS SECONDARY ENDPOINT SELECTION OF SPECIMENS SPECIMENS AND SUBJECTS PROVIDING SPECIMENS 6.1.1 Subject Screening 6.1.2 Informed Consent 6.1.2.1 Special Circumstances for Informed Consent ELIGIBILITY CRITERIA | 19<br>19<br>20<br>20<br>20<br>21<br>21<br>21 |
| 5.<br>5.1<br>5.2<br>6.<br>6.1 | ENDPOINTS PRIMARY ENDPOINTS SECONDARY ENDPOINT SELECTION OF SPECIMENS SPECIMENS AND SUBJECTS PROVIDING SPECIMENS 6.1.1 Subject Screening 6.1.2 Informed Consent 6.1.2.1 Special Circumstances for Informed Consent ELIGIBILITY CRITERIA 6.2.1 Inclusion Criteria 6.2.2 Exclusion Criteria | 19<br>19<br>20<br>20<br>20<br>21<br>21<br>21<br>21<br>22 |
| 5.<br>5.1<br>5.2<br>6.<br>6.1 | ENDPOINTS | 19<br>19<br>20<br>20<br>20<br>21<br>21<br>21<br>21<br>22<br>22 |
| 5.<br>5.1<br>5.2<br>6.<br>6.1 | ENDPOINTS | 19<br>19<br>20<br>20<br>20<br>21<br>21<br>21<br>21<br>22<br>22 |




| | 7.1.1 | Adverse Event | 23 |
|---|---|---|---|
| | 7.1.2 | Serious Adverse Event | 23 |
| | 7.1.3 | Device Deficiency/Device Malfunction | 23 |
| 7.2 | DEVIC | RELATIONSHIP | 24 |
| | 7.2.1 | Unanticipated (Serious Adverse) Device Effect [U(S)ADE] | 24 |
| 7.3 | ADVER | SE EVENT AND DEVICE DEFICIENCY/DEVICE MALFUNCTION REPORTING | 24 |
| | | Adverse Event Reporting | |
| | | Unanticipated Serious Adverse Device Effect Reporting to Sponsor and EC | |
| | | Device Deficiency/Malfunction Reporting | |
| _ | | | |
| | | | ä |
| _ | | | |
| = | | | |
| _ | | | |
| = | | | |
| 9.2 | FINAN | CES AND AGREEMENTS | 20 |
| _ | 1 1147-114 | JEO AND ACKEEMENTO | 20 |
| 9.4 | TRAIN | NG | 29 |
| | 9.4.1 | Site Training | 29 |
| 9.5 | MONIT | ORING | 29 |
| 9.6 | DEVIA | TIONS FROM CPSP | 30 |
| _ | | | |






| 32<br>32 |
|----------|
| 33<br>33 |
| 35 |
| 36 |
| 37<br>37 |
| 38 |
| _ |



#### 1. INTRODUCTION

Rapid antigen detection (RAD) tests are used to perform rapid diagnosis of SARS-CoV-2 infection based on a qualitative approach. RAD tests detect the viral antigen by the immobilized coated SARS-CoV-2 antibody placed on the device. The results of these tests are available in a short time, reducing the workload in diagnostic hospitals and laboratories and improving the turn-around time.

EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test is an *in vitro* Diagnostic (IVD) medical device intended to be used for the qualitative detection of SARS-CoV-2 nucleocapsid antigen. The result from this IVD test identifies the presence or absence of the SARS-CoV-2 antigen as an aid for the diagnosis of COVID-19 infection.

#### 1.1 Background and rationale

In 2019 a novel corona virus, designated as SARS-CoV-2 and associated with unusual viral pneumonia named Corona virus Disease 19 (COVID-19), sprouted in the city of Wuhan, China, and rapidly spread to create a global pandemic. Identification of people infected with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is essential for controlling its spreading and public health management.

Since the beginning of the COVID-19 outbreak, tests that can enable both mass screening and reliable detection of infected people are needed<sup>1</sup>. The reliance on testing underscores the importance of analytical sensitivity of virus assays, being the real-time quantitative polymerase chain reaction (RT-qPCR) from nasopharynx swab the gold-standard <sup>2</sup>. However, RT-PCR is expensive, time-consuming, and requires specialized laboratory personnel and instrumentation compared to rapid tests <sup>3</sup>.

New developments in SARS-CoV-2 diagnostics have the potential to reduce cost and turnaround time <sup>4-6</sup>. Several diagnostic strategies are available for identifying or ruling out current infection, identifying people in need of care escalation, or testing for past infection and immune response. Point-of-care (POC) antigen and molecular tests for the detection of current SARS-CoV-2 infections are rapid antigen detection (RAD) tests, which allow earlier detection and isolation of confirmed cases compared to laboratory-based diagnostic methods.

Coronavirus RAD tests, have demonstrated good sensitivity and specificity in comparison to RT-qPCR <sup>7-9</sup>. Moreover, previous studies have shown that RADs can exhibit high sensitivity in detecting samples containing infectious virus, indicating a high sensitivity to detect contagious individuals <sup>10,11</sup>

The RAD tests, based on the immunochromatographic principle, detect SARS-CoV-2 nucleocapsid protein (N)

| t or near the place where a specimen is collected, providing results within few minutes <sup>3</sup> . In general, RAD tests<br>onsist of fixing match-paired antibodies to the surface of the cassette and coupling an anti-antigen match- |
|---|
| aired antibodies to the detection nanoparticles. |
| uGeni SARS-CoV-2 Ag RDT is a fluorescent immunochromatographic RAD test for COVID-19 rapid detection |
| sing the state of |
| rovide positive, negative, or invalid result for the presence of SARS-CoV-2 antigen. The EuGeni device is |
| tended to be used by healthcare professionals only |

Template CA-06.17.02-A 



#### 2. IN-VITRO DIAGNOSTIC MEDICAL DEVICE OVERVIEW

#### 2.1 IVD Medical Device under investigation






#### 2.3 Intended User

for internal assay control.

The EuGeni SARS-CoV-2 Ag RDT is intended to be used by healthcare professionals which must be qualified and trained. This test is intended for use at the Point of Care (POC) and laboratory settings.

# 2.4 Mechanism of action of the Device Under Investigation The EuGeni SARS-CoV-2 Ag RDT is a test strip based on lateral flow technology for detection but not differentiation of SARS-CoV and SARS-CoV-2 antigen, and

The test line contains an immobilized monoclonal mouse antibody to capture SARS-CoV-2 antigen and the control line contains an immobilized control anti-mouse antibody

| control line contains a | an immobilized control anti-mouse antibody. |
|---|---|
| • | |
| | The control line must be detected by the |
| | for the test to be valid. If the control line is not detected, the test is considered invalid |

and must be repeated using another test cassette.

For more precise information on the device description and the reader, please refer to the IFU.

#### 2.5 Device Handling

All investigational products shall be stored according to the labeling and Instructions for Use (IFU) in a secure area to prevent unauthorized access or use.

| <u> </u> |
|----------|

For further device handling warnings and precautions, please see the details in the IFU.




#### 3. CLINICAL PERFORMANCE STUDY OVERVIEW

#### 3.1 Clinical Performance study Objective

The objective of this clinical performance study (CPS) is to determine the diagnostic accuracy (sensitivity and specificity) of the EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test in the diagnosis of SARS-CoV-2 in specimens from subjects suspected of COVID-19 disease or with unknown COVID-19 status.




#### 4. CLINICAL PERFORMANCE STUDY DESIGN AND PROCEDURES

#### 4.1 Clinical performance study design

This clinical performance study (CPS) is designed as a non-interventional, two-arm, prospective, non-randomized, open-label and multi-center study. The two study arms as defined depending on the specimen collection method:

- 1. Nasopharyngeal specimen collection for comparison with gold-standard RT-PCR
- Combined nasal mid-turbinate and throat specimen collection for comparison with gold-standard RT-PCR

The expected minimum number of specimens for this CPS is 1850, divided as follows:

Nasopharyngeal specimen collection:

| • | 300 positive specimens collected from subjects at different timepoints post onset of symptoms: |
|---|---|

- 120 negative specimens from hospitalized patients
- 505 negative specimens from subjects with respiratory symptoms

Combined nasal mid-turbinate and throat specimen collection:

| • | 300 positive specimens collected from subjects at different timepoints post onset of symptoms: 120 negative specimens from hospitalized patients 505 negative specimens from subjects with respiratory symptoms. |
|---|---|
| • | |
| | The estimated numbers for each nen type are approximate and may vary depending on the natural recruitment at the investigational sites are the correct distribution of sample size requirements. |
| or the | udy has been designed to involve as little pain, discomfort, fear and any other foreseeable risk as possible subjects, and both the risk threshold and the degree of distress are specifically defined in the clinical nance study plan (CPSP) and constantly monitored. |
| | PS will be conducted in up to 10 sites in Europe. The primary and secondary endpoints will be evaluated all specimens have been collected and analyzed. |

#### 4.2 Clinical Performance Study Procedures

The Clinical Performance Study will occur in a single subject visit, and no clinical follow up will be required.

#### 4.2.1 Informed Consent and Specimen collection

Before starting any study-related activity, the subject must have provided the signed informed consent form following the requirements in [Section 6.1.2]. Next, the specimen collection will be performed by professionally trained and qualified healthcare personnel.






Rapid Diagnostic Test IFU.

One bilateral swab will be taken to be analyzed with the device under investigation and another bilateral swab will be taken to be analyzed with the gold-standard RT-PCR. The specimen collection method for EuGeni analysis will be performed using either a combined nasal mid-turbinate and throat swab, or a nasopharyngeal swab, which will determine the inclusion into one of the two study arms. Enrolment into the combined nasal mid-turbinate and throat arm or nasopharyngeal will not be randomized, however consecutive and parallel enrollment in both arms will take place. Regardless of the study arm, the RT-PCR specimen collection will always occur to allow result comparison between the investigational device and RT-PCR.

| always occur to allow result comparison between the investigational device ar | id RT-PCR. |
|---|---|
| For further information on specimen collection, please refer to IFU | |
| 4.2.2 Specimen analysis procedure | |
| The specimen analysis shall be performed by professional healthcare personne the gold-standard RT-PCR shall follow the procedures established by the standard RT-PCR shall follow the procedures established the procedures are standard RT-PCR shall follow the procedures established the procedures are standard RT-PCR shall follow the procedures are stan | 이 아이지 않는 그리다 이 아이를 잃었는 아이지는 그러워 하는 것이 되었다. 그런데 되었다면 모양하다 되었다. |
| Those specimens analyzed by the EuGeni SARS-CoV-2 Antigen Rapid I procedures laid down in the IFU and protocol. | Diagnostic Test shall follow the |
| a) Positive results indicate the presence of SARS-CoV-2-antigen and is 2 infection. | indicative of primary SARS-CoV- |
| b) Negative results indicate the specimen does not contain SARS-CoV control line will be displayed. Negative results should be tronot be used as the sole basis for clinical diagnosis and treatment. | |
| c) If a test is Invalid, a new test should be performed with a new subject | ot specimen and a new cassette. |
| For more information on the interpretation of results, please refer to the | ne EuGeni SARS-CoV-2 Antiaen |






All results obtained from the investigational device should only be noted in the Case Report Form. These results will not impact or drive patient management decisions. The gold-standard RT-PCR results will provide this information to the healthcare professionals and the enrolled subjects.

#### 4.2.2.1 Specimen handling and storage

Template CA-06.17.02-A






#### 4.3 Measures Taken to Avoid and Minimize Bias

This clinical performance study has been designed to be multicenter in order to minimize bias related to site specific standard of care patient and specimen collection method.

All participants who meet the inclusion and exclusion criteria will be eligible to join the study. Inclusion into the two study arms will not be randomized, however sites will be instructed to consecutively enroll subjects into both arms. Recruitment at each investigational site will be limited to of the total sample size.

To avoid bias related to the collection method, all study subjects will have a bilateral swab specimen collection for investigational device analysis and for RT-PCR analysis, for direct comparison within the same subjects.

#### 5. ENDPOINTS

#### 5.1 Primary Endpoints

The primary endpoint of this clinical performance study is to assess the EuGeni SARS-CoV-2 Ag RDT diagnostic accuracy in terms of sensitivity and specificity measured as the following:

- The diagnostic sensitivity of EuGeni SARS-CoV-2 Ag RDT, defined as the ability to identify the presence
  of a target marker associated with SARS-CoV-2, of nasopharyngeal specimens and combined nasal
  mid-turbinate and throat specimens, respectively, compared with gold-standard SARS-CoV-2 RT-PCR.
- The diagnostic specificity of EuGeni SARS-CoV-2 Ag RDT, defined as the ability to recognise the
  absence of a target marker associated with SARS CoV-2, of nasopharyngeal specimens and combined
  nasal mid-turbinate and throat specimens, respectively, compared with gold-standard SARS-CoV-2 RTPCR.

#### 5.2 Secondary Endpoint

The secondary endpoint of this clinical performance study is to compare the EuGeni SARS-CoV-2 Ag RDT diagnostic accuracy (specificity and sensitivity) between the two specimen collection methods (nasopharyngeal and combined nasal mid-turbinate and throat) to assess any potential impact on diagnostic accuracy.




#### 6. SELECTION OF SPECIMENS

#### 6.1 Specimens and subjects providing specimens

The specimens used in this clinical performance study will be selected from any gender of subjects of the general population suspected to be infected with SARS-CoV-2 or with unknown COVID-19 status.

The Principal Investigator or designee, previously trained in this CPSP, will revise subject and specimen eligibility according to the inclusion/exclusion criteria. Those who meet all the inclusion criteria and no exclusion criteria shall be suitable to participate in the study.

#### 6.1.1 Subject Screening

Enrolled subjects will be fully informed about the clinical performance study, following the established Informed Consent process (described in the next section). Once a duly dated and signed Informed Consent form is obtained, the clinical performance procedures may begin. Subjects under 18 years of age must be accompanied by a parent or legal representative who must also give consent for the under-age's participation in the study.

| • |
|---|
| In case the subject does not meet all inclusion criteria or meets any of the exclusion criteria, the subject is considered a screening failure. The Principal Investigator or the delegated clinical performance study personnel will record the screening failure in the hospital records and on the screening log as required. |
| Subjects meeting general inclusion criteria and no exclusion criteria will be asked to sign an Informed Consent form if they wish to participate in the clinical performance study. |
| Subject data will be collected following enrollment into the clinical performance study. |
| 6.1.2 <u>Informed Consent</u> |
| The Investigator or his/her authorized designee (if applicable) will conduct the Informed Consent process, as required by applicable regulations and the center's EC. |
| Withdrawal from the clinical performance study will not jeopardize their future medical care or relationship with the investigator. |
| During the discussion, the Principal Investigator or his/her authorized designee will avoid any improper influence on the subject and will respect subject's legal rights. Financial incentives will not be given to the subject. |
| The subject shall have adequate time to review, ask questions, and consider participation. |
| quodiono, ana conolaci participation. |


Template CA-06.17.02-A






| If the subject agrees to participate, the Informed |
|---|
| Consent form must be signed and dated by the subject and thereafter by the person obtaining the consent prior |
| to any clinical performance study-specific procedures. |

#### 6.1.2.1 Special Circumstances for Informed Consent

#### Individuals under age of 18 or under age of legal consent:

Individuals who are minors (under the age of 18 or age of legal consent, but over 12 years old) may be enrolled in this clinical performance study. Informed consent must be obtained using the IRB/EC approved informed consent in accordance with IRB/EC requirements.

In this special circumstance, the legally acceptable representative will represent the individual during the Informed Consent process, which will be performed according to the requirements in [Section 6.1.2]. The minor will also be informed about the CPS within his/her ability to understand.

#### 6.2 Eligibility Criteria

#### 6.2.1 Inclusion Criteria

- Specimens from subjects over 12 years old agreeing to participate in the study and with a legal representative able to provide informed consent, OR;
- 2. Specimens from subjects over 18 years old able to provide informed consent.
- Specimens collected with nasopharyngeal swabs, OR;
- 4. Combined nasal mid-turbinate and throat specimens' collection.

#### 6.2.2 Exclusion Criteria

- Specimens and testing methods that are deemed not compatible with gold-standard RT-PCR standards.
- 2. Specimens stored for over 2 hours at 2-8 °C in between collection and testing with EuGeni SARS-CoV-2 Ag RDT
- 3. Specimens stored for over 5 days at -20°C between collection and testing with RT-PCR.
- 4. Specimens stored for over 24h at 4°C between collection and testing with RT-PCR.
- 5. Contamination and/or deterioration of the specimen which, in the opinion of the investigator, may affect its handling and/or analysis.
- 6. The subject is deemed unsuitable to participate in the study by the investigator.






#### 6.3 Subject Enrolment

A subject is considered enrolled in the CPS from the moment the subject provides written informed consent and has been confirmed to meet all inclusion criteria and none of the exclusion criteria.

| • |
|---|

#### 6.4.1 Suspension or Early Termination of the Clinical Performance Study

While no formal statistical rule for early termination of the clinical performance study for insufficient accuracy of the device under investigation is defined, the Sponsor reserves the right to discontinue the clinical performance study at any stage with suitable written notice to the investigator. Possible reason(s) may include, but are not limited to:

- Unanticipated adverse device effect (e.g., UADE) occurs and it presents an unreasonable risk to the participating subjects.
- · Further product development is cancelled.

| Should the clinical performance study be di hospital practice with device-related AEs requirements. | reported to the Sponso | |
|---|---|---|
| | | 2 |




#### 7. ADVERSE EVENTS

| he study has been designed to involve as little pain, discomfort, fear, and any other foreseeable risk as possibl |
|---|
| or subjects. |

#### 7.1 Definition

#### 7.1.1 Adverse Event

An adverse event (AE) is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device under investigation.

Note 1: This definition includes events related to the medical device under investigation or the comparator.

Note 2: This definition includes events related to the procedures involved.

**Note 3:** For users or other persons, this definition is restricted to events related to medical devices under investigation.

#### 7.1.2 Serious Adverse Event

If the AE meets any of the criteria below, it is regarded as a serious adverse event (SAE).

- a) Led to a death,
- b) Led to a serious deterioration in health of the subject, that either resulted in
  - 1. a life-threatening illness or injury, or
  - 2. a permanent impairment of a body structure or a body function, or
  - 3. in-patient hospitalization or prolongation of existing hospitalization, or
  - 4. medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.
  - 5. chronic disease
- c) Led to fetal distress, fetal death or a congenital abnormality or birth defect.

**Note:** A planned hospitalization for pre-existing condition, or a procedure required by the CIP, without a serious deterioration in health, is not considered to be an SAE.

#### 7.1.3 Device Deficiency/Device Malfunction

Device deficiency is defined as an inadequacy of a medical device related to its identity, quality, durability, reliability, safety or performance, such as malfunction, misuse or use error and inadequate labeling. This includes the failure of the device to meet its performance specifications or otherwise perform as intended. Note: Performance specifications include all claims made in the labeling of the device.

Template CA-06.17.02-A 



A device malfunction is the failure of a device to meet its performance specifications or otherwise perform as intended, when used in accordance with the instructions for use or CPSP.

#### 7.2 Device Relationship

Determination of whether there is a reasonable possibility that an investigational product or device under investigation caused or contributed to an AE is to be performed by the Investigator and recorded on the appropriate CRF form. Determination should be based on assessment of temporal relationships, evidence of alternative etiology, medical/biologic plausibility, and patient condition (pre-existing condition).

#### 7.2.1 Unanticipated (Serious Adverse) Device Effect [U(S)ADE]

Unanticipated serious adverse device effect (USADE) refers to any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.

#### 7.3 Adverse Event and Device Deficiency/Device Malfunction Reporting

#### 7.3.1 Adverse Event Reporting

# General AE Reporting

| All adverse event | data, |
|---|---|
| | will be reported to the Sponsor on a |
| CRF. Additional information with regard to an adverse | e event should be updated within the appropriate CRF. |
| Unchanged, chronic, non-worsening or pre-existing c | onditions are not AEs and should not be reported. |

All adverse events will be collected on each subject through the study duration

#### SAE Reporting

The investigator should report all SAEs to the Sponsor as soon as possible but no later than outlined below.

| Clinical Site | Reporting timelines |
|---|---|
| All Sites | SAEs must be reported to the Sponsor no later than 3 calendar days from the day the site personnel became aware of the event |






#### 7.3.2 <u>Unanticipated Serious Adverse Device Effect Reporting to Sponsor and EC</u>

The Sponsor requires the Investigator to report any USADE to the Sponsor within 3 calendar days of the investigator's knowledge of the event,

#### 7.3.3 <u>Device Deficiency/Malfunction Reporting</u>

All device deficiencies/malfunctions should be reported on the appropriate CRF form.

The investigator should report all device deficiencies/malfunctions to the Sponsor as soon as possible but no later than outlined below.

| Clinical Sites | Reporting timelines |
|---|---|
| All Sites | Device deficiencies/malfunctions must be reported to the Sponsor no later than 3 calendar days from the day the site personnel became aware of the event |






| 8. | STATISTICAL CONSIDERATIONS |
|---|---|
| Ξ | |
| | 8.1 Analysis Populations |
| Ξ | |
| | <ul> <li>Arm 1, including specimens collected with nasopharyngeal swabs</li> <li>Arm 2, including specimens collected with combined nasal mid-turbinate and throat swabs</li> <li>8.2 <u>Statistical Analyses</u></li> </ul> |

#### 8.2.1 Primary Diagnostic Accuracy Endpoint(s) Analyses

The evaluation of the accuracy of the EuGeni SARS-CoV-2 Ag RDT in the diagnosis of COVID-19 will be analyzed by means of the sensitivity and specificity capacity of this test.






# 8.2.2 Secondary Endpoint Analysis The secondary endpoint assesses any potential impact of the specimen collection method (arms 1 and 2) on EuGeni SARS-CoV-2 Ag RDT diagnostic accuracy (specificity and sensitivity rates). 8.3 Sample Size Calculation and Assumptions The sample size calculation is based on the objective to demonstrate an 80% sensitivity and a 98% specificity

| 8.3 Sample Size Calculation and Assumptions |
|---|
| The sample size calculation is based on the objective to demonstrate an 80% sensitivity and a 98% specificing the Figure 200 MP 40 to the first sensitivity and a 98% specificing the Figure 200 MP 40 to the first sensitivity and a 98% specificing the Figure 200 MP 40 to the first sensitivity and a 98% specificing the Figure 200 MP 40 to the first sensitivity and a 98% specificing the first sensitivity and a 98% specifical sensitivity and a 98% spec |
| of the EuGeni SARS-CoV-2 Ag RDT for COVID-19 testing, |






| | 6 |
|---|---|
| W | |
| 7 | |




#### 9. QUALITY CONTROL AND QUALITY ASSURANCE

| 9.1 <u>Selection of Clinical Sites and Investigators</u> | |
|---|---|
| The Sponsor or designee will select investigators qualified by education, training and experience to participating the clinical performance study. | ate |
| in the similar perfermance study. | |
| 9.2 Finances and Agreements | |
| The clinical performance study will be financed by AnteoTech., Ltd. | |
| <u> </u> | _ |
| 9.4 <u>Training</u> | |
| 9.4.1 Site Training | |
| All Investigators and clinical performance study personnel are required to attend Sponsor training session which may be conducted at an Investigator's meeting, a site initiation visit, or other appropriate training session | |
| Video call or self-training may take place as required. | |
| 9.5 Monitoring | |
| Sponsor and/or designee will monitor the clinical performance study over its duration according to the CPS specific monitoring plan which will include the planned extent of source data verification. This monitoring plan will be a separate document that can be updated during the course of the study. | |




AnteoTech LTD.
EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test
Clinical Performance Study
CPSP Ver 3.0, 19Sep2022

| 9.6 <u>Deviations from CPSP</u> The Investigator should not deviate from the CPSP for any reason except in cases of medical emergencia when the deviation is necessary to protect the rights, safety and well-being of the subject or eliminate apparent immediate hazard to the subject. In that event, the Investigator will notify Sponsor immediately liphone or in writing. |
|---|






| • |
|-----------------------------------------|
| ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, |
| _ |




AnteoTech LTD.
EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test
Clinical Performance Study
CPSP Ver 3.0, 19Sep2022

| 10.1 Protection of Personally Identifiable Information The Sponsor respects and protects personally identifiable information collected or maintained for this clinical performance study. |
|---|
| The Sponsor requires the investigational sites to transfer into Sponsor's data management systems only pseudonymous Personal Information (key-coded) necessary to conduct the clinical performance study, such as the patient's medical condition, treatment, dates of treatment, etc. |

The Sponsor maintains a Privacy Incident procedure that complies in all respects with Applicable Law and industry best practices.

#### 10.2 Data Management Plan

Template CA-06.17.02-A

A Data Management Plan (DMP) will describe procedures used for data entry and collection. Data review and data cleaning, and issuing, resolving data discrepancies and methods for data base lock.






| 10.4 Case Report Form Completion |
|---|
| Primary data collection based on source-documented hospital and/or clinic chart reviews will be performed clearly and accurately by site personnel trained on the CPSP and CRF completion. |

#### 10.5 Record Retention

The Sponsor and Investigator/Site will archive and retain all documents pertaining to the CPS as per the applicable regulatory record retention requirements. The Investigator must obtain permission from Sponsor in writing before destroying or transferring control of any CPS records.









#### 11. RISK ANALYSIS

Recruited subjects for specimen collection may have anticipated risks associated with the specimen collection procedure. A risk analysis is conducted and identified risks are similar to those well-known for standard of care collection procedures (e.g., swab collection for gold-standard RT-PCR) and are described in the IFU.

| 8 | |
|---|----|
| | 99 |
| | 9 |
| | Ţ |




#### 11.6 Benefit to Risk Rationale

While there are no additional risks associated with study participation, the public health may be benefitted.






#### 12. ETHICAL CONSIDERATION

#### 12.1 Institutional Review Board/Ethics Committee Review and Approval

| Institutional | Review | Board | (IRB)/Ethics | Committee | (EC) | approval | for | the | CPSP | and | ICF/other | writter |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| information | provided | to the p | atient will be | obtained at e | each ir | rvestigatio | nal s | site p | rior to c | onse | nting and e | nrolling |
| patients in t | his clinica | al perfor | mance study. | The approv | al lette | er must be | rece | eived | prior to | the s | start of this | clinical |
| performance | e study a | nd a co | py must be pr | ovided to the | Spor | nsor. | | | | | | |
| | .40* | | | | | | | | | | | |

| y | |
|---|--------|
| | - 1 |
| | <br>r. |




#### 13. CLINICAL PERFORMANCE STUDY CONCLUSION

The clinical performance study will be concluded when:

- · The investigational site is closed AND
- The final report has been provided to investigators or the Sponsor has provided formal documentation of clinical performance study closure.

The Sponsor shall submit the clinical performance study report (CPSR) within one year of the end of the investigation as applicable per the study.




AnteoTech LTD. EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test Clinical Performance Study CPSP Ver 3.0, 19Sep2022

| 14. | PUBL | ICATION | N POLICY |
|-----|------|---------|----------|

| The data and results from the clinical performance study are the sole property of the Sponsor. |
|---|




#### **APPENDIX I: ABBREVIATIONS AND ACRONYMS**

| Abbreviation/Acronym | Words |
|----------------------|-------------------------------------|
| AE | Adverse Event |
| ADE | Adverse Device Effect |
| CPS | Clinical Performance Study |
| CPSP | Clinical Performance Study Plan |
| CPSR | Clinical Performance Study Report |
| CRF | Case Report Form |
| СТА | Clinical Trial Agreement |
| DMP | Data Management Plan |
| EC | Ethics Committee |
| EDC | Electronic Data Capture |
| ICF | Informed Consent Form |
| IFU | Instructions For Use |
| IVD | In vitro Diagnostic |
| RT-PCR | Real-Time Polymerase Chain Reaction |
| PI | Principal Investigator |
| RAD | Rapid Antigen Detection |
| RDT | Rapid Diagnostic Test |
| SAP | Statistical Analysis Plan |
| SAE | Serious Adverse event |












| • | |
|---|----------|
| • | |
| • | |
| _ | |
| • | |
| _ | · |
| | <u> </u> |










